CLINICAL TRIAL: NCT03998254
Title: A Phase 3 Randomized, Double-Blinded, Controlled With GARDASIL® Efficacy, Immunogenicity and Safety Study of V503 [a 9-Valent HPV Vaccine] in Chinese Women 20 to 45 Years of Age
Brief Title: Efficacy, Immunogenicity and Safety of V503 in Chinese Women Aged 20-45 Years (V503-023)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V503-023; V503-023 (Other: Merck)
Record Dates: First submitted 2019-06-21; First posted 2019-06-26 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- V503 (Experimental): Single 0.5-mL intramuscular injection at Day 1, Month 2, and Month 6
  Interventions: Drug: V503
- Gardasil (Active Comparator): Single 0.5-mL intramuscular injection at Day 1, Month 2, and Month 6
  Interventions: Drug: Gardasil

INTERVENTIONS:
Drug: V503 — 9vHPV [Types 6, 11, 16, 18, 31, 33, 45, 52, and 58] L1 virus-like particle vaccine
  Arms: V503
Drug: Gardasil — qHPV [Types 6, 11, 16, and 18] L1 virus-like particle vaccine
  Arms: Gardasil

SUMMARY:
This study will evaluate the efficacy, immunogenicity and safety of 9-valent human papillomavirus (9vHPV; V503) vaccine in Chinese women 20 to 45 years of age. The primary hypotheses are: 9vHPV vaccine reduces the incidence of HPV 31-, 33-, 45-, 52-, and 58-related 12-month persistent infection at least 1 month post Dose 3, compared with quadrivalent HPV (qHPV) vaccine in women 20 to 45 years of age who are seronegative at Day 1 and polymerase chain reaction (PCR) negative Day 1 through Month 7 to the relevant HPV type; and 9vHPV vaccine induces non-inferior competitive luminex immunoassay (cLIA) geometric mean titers (GMTs) for each of HPV 6, 11, 16, and 18 one month post Dose 3, compared with qHPV vaccine in women 20 to 45 years of age who are seronegative at Day 1 and PCR negative Day 1 through Month 7 to the relevant HPV type.

DETAILED DESCRIPTION:
This study has two stages with the Stage I expected from Day 1 through Month 30, and the Stage II expected post-Month 30 to Month 90. The Stage I study is a case-driven study which aims to accrue at least 20 cases of HPV 31/33/45/52/58-related 12-month persistent infection and at least 39 cases of HPV 31/33/45/52/58-related 6-month persistent infection by completion of Month 30 visit. The Stage II study is a case-driven study which aims to accrue at least 12 cases of HPV 31/33/45/52/58-related cervical intraepithelial neoplasia grade 2 or 3 (CIN 2/3), cervical adenocarcinoma in situ (AIS), and cervical cancer observed in both Stage I and Stage II, by completion of Month 90 visit.

ELIGIBILITY:
Inclusion Criteria

* Healthy
* Has not had sex with males or has had sex with males and used effective contraception with no failures since the first day of the participant's last menstrual period through Day 1
* Agrees to use effective contraception if has sex with a male partner during study
* Has had sexual intercourse with male partners, and has had 1 to 4 male and/or female sexual partners

Exclusion Criteria

* History of a positive test for HPV
* History of an abnormal Pap test result showing ASC-US, atypical squamous cells - cannot exclude HSIL (high grade squamous intraepithelial lesion [(ASC-H)], low-grade squamous intraepithelial lesion (LSIL), HSIL), or atypical glandular cells
* History of an abnormal cervical biopsy result showing CIN, adenocarcinoma in situ or cervical cancer
* History of or clinical evidence at the Day 1 gynecologic examination of HPV-related anogenital diseases (e.g., genital warts, VIN, VaIN, AIN, vulvular cancer, vaginal cancer or anal cancer
* Does not have an intact cervix uteri or has more than one cervix uteri
* Is pregnant
* Known allergy to any vaccine component, including aluminum, yeast, or Benzonase™ (nuclease, Nycomed™ [used to remove residual nucleic acids from this and other vaccines])
* History of severe allergic reaction (e.g., swelling of the mouth and throat, difficulty breathing, hypotension or shock) that required medical intervention
* Has thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injections
* Currently immunocompromised or has been diagnosed as having a congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease, or other autoimmune condition
* Has had a splenectomy
* Is expecting to donate eggs during Day 1 through Month 7 of the study
* Plans to receive during Day 1 through Month 7 of the study, is receiving or has received within 12 months prior to enrollment the following immunosuppressive therapies: radiation therapy, cyclophosphamide, azathioprine, methotrexate, any chemotherapy, cyclosporin, leflunomide (Arava™), tumor necrosis factor (TNF)-α antagonists, monocolonal antibody therapies (including rituximab [Rituxan™]), intravenous gamma globulin (IVIG), antilymphocyte sera, or other therapy known to interfere with the immune response. With regard to systemic corticosteroids, a participant will be excluded if she is currently receiving steroid therapy, has recently (defined as within 2 weeks of enrollment) received such therapy, or has received 2 or more courses of high dose corticosteroids (orally or parenterally) lasting at least 1 week within 12 months prior to enrollment. Participants using inhaled, nasal, or topical corticosteroids are considered eligible for the study.
* Plans to receive during Day 1 through Month 7 of the study, is receiving or has received within the 6 months prior to the Day 1 vaccination any immune globulin product (including RhoGAM™) or blood derived product other than IVIG
* Has received a marketed HPV vaccine, or has participated in an HPV vaccine clinical study and has received either active agent or placebo
* Concurrently enrolled in clinical studies of investigational agents or studies involving collection of cervical specimens
* User of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence at the discretion of the investigator. Alcohol abusers are defined as those who drink despite recurrent social, interpersonal, and/or legal problems as a result of alcohol use

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only females will be enrolled
Enrollment: 6000 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Stage I: Combined Incidence of HPV 31-, 33-, 45-, 52-, and 58-related 12-month Persistent Infection | 1 month post vaccination 3 (Month 7) up to Month 30
  A 12-month persistent infection This endpoint is defined to have occurred if a participant who is positive for the same HPV type by the HPV PCR assay in the LVPP/EEC swabs, biopsy, ECC or definitive therapy samples obtained in 3 or more consecutive visits over a period of at least 12 months. Incidence is defined as the number of cases of persistent infection per 10,000 person-years of follow-up in a treatment arm.
Stage I: Geometric Mean Titers to HPV Types 6, 11, 16, and 18 Antibodies | 1-month post vaccination 3 (Month 7)
  Serum antibodies to HPV types 6/11/16/18 are measured with a Competitive Luminex Immunoassay (cLIA). Titers are reported in milli Merck Units/mL.
Stage I: Percentage of Participants Who Report at Least 1 Solicited Injection-site Adverse Event | up to 8 days post any vaccination
  An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study vaccine or protocol-specified procedure is also an AE. AEs such as redness, swelling, and pain/tenderness/soreness at the injection site are recorded.
Stage I: Percentage of Participants Who Report at Least 1 Solicited Systemic Adverse Event | up to 30 days post any vaccination
  An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study vaccine or protocol-specified procedure is also an AE. Systemic AEs are those not categorized as injection-site AEs.
Stage I: Percentage of Participants Who Experience at Least 1 Serious Adverse Event (SAE) | Day 1 up to approximately Month 30
  An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study vaccine or protocol-specified procedure is also an AE. An SAE is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, or is another important medical event.
Stage II: Combined Incidence of HPV 31-, 33-, 45-, 52-, and 58-related CIN 2/3, AIS, and cervical cancer | Month 7 up to Month 90
  This endpoint is defined to have occurred if on a single cervical biopsy, ECC, LEEP or Conization (cold knife/laser) specimen, there is: (a) a HPV Pathology Panel consensus diagnosis of CIN (grade 2 or 3), AIS, or cervical cancer; AND (b) detection of at least 1 of HPV types 31, 33, 45, 52 or 58 by Thinsection PCR in an adjacent section from the same tissue block. Disease incidence is defined as the number cases per 10,000 person-years of follow-up in a treatment arm.
Stages I/II: Percentage of Participants Who Experience at Least 1 Serious Adverse Event (SAE) | Day 1 up to approximately Month 90
  An AE is defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with study vaccine. An AE can therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of study vaccine or a protocol-specified procedure, whether or not considered related to the study vaccine or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the study vaccine or protocol-specified procedure is also an AE. An SAE is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, or is another important medical event.

SECONDARY OUTCOMES:
Stage I: Combined Incidence of HPV 31-, 33-, 45-, 52-, and 58-related 6-month Persistent Infection | 1 month post vaccination 3 (Month 7) up to Month 30
  A 6-month persistent infection is defined to have occurred if a participant who is positive for the same HPV type by the HPV PCR assay in the LVPP/EEC swabs, biopsy, ECC or definitive therapy obtained in 2 or more consecutive visits over a period of at least 6 months. Incidence is defined as the number of cases of persistent infection per 10,000 person-years of follow-up in a treatment arm.
Stage I: Percentage of Participants Who Seroconvert by cLIA to HPV Types 6, 11, 16, and 18 | 1 Month Post Vaccination 3 (Month 7)
  Serum antibody titers for HPV types 6, 11, 16, and 18 will be determined using cLIA. The percentage of participants that achieve the serostatus cut-offs for seroconversion for each HPV type will be summarized.
Stage I: Combined Incidence of HPV 31-, 33-, 45-, 52-, and 58-related 12-month Persistent Cervical Infection | 1 month post vaccination 3 (Month 7) up to Month 30
  A 12-month persistent cervical infection is defined to have occurred if a participant who is positive for the same HPV type by the HPV PCR assay in the EEC swabs, cervical biopsy, ECC or cervical definitive therapy samples obtained in 3 or more consecutive visits over a period of at least 12 months. Incidence is defined as the number of cases of persistent infection per 10,000 person-years of follow-up in a treatment arm.
Stage I: Combined Incidence of HPV 31-, 33-, 45-, 52-, and 58-related 12-month Persistent Non-cervical Infection | 1 month post vaccination 3 (Month 7) up to Month 30
  A 12-month persistent non-cervical infection is defined to have occurred if a participant who is positive for the same HPV type by the HPV PCR assay in the LVPP swabs, biopsy, or definitive therapy samples obtained from the external genitalia in 3 or more consecutive visits over a period of at least 12 months. Incidence is defined as the number of cases of persistent infection per 10,000 person-years of follow-up in a treatment arm.
Stage I: Combined Incidence of HPV 31-, 33-, 45-, 52-, and 58-related 6-month Persistent Cervical Infection | 1 month post vaccination 3 (Month 7) up to Month 30
  A 6-month persistent cervical infection is defined to have occurred if a participant who is positive for the same HPV type by the HPV PCR assay in the EEC swabs, cervical biopsy, ECC or cervical definitive therapy samples obtained in 2 or more consecutive visits over a period of at least 6 months. . Incidence is defined as the number of cases of persistent infection per 10,000 person-years of follow-up in a treatment arm.
Stage I: Combined Incidence of HPV 31-, 33-, 45-, 52-, and 58-related 6-month Persistent Non-cervical Infection | 1 month post vaccination 3 (Month 7) up to Month 30
  A 6-month persistent non-cervical infection is defined to have occurred if a participant who is positive for the same HPV type by the HPV PCR assay in the LVPP swabs, biopsy, or definitive therapy samples obtained from the external genitalia in 2 or more consecutive visits over a period of at least 6 months. . Incidence is defined as the number of cases of persistent infection per 10,000 person-years of follow-up in a treatment arm.
Stage I: Combined Incidence of Papanicolaou (Pap) Test Abnormalities That are Related to HPV 31, 33, 45, 52, or 58 | Month 7 up to Month 30
  This endpoint is defined to have occurred if a participant is found to have: (a) a Pap test result of ASC-US positive for high risk HPV, LSIL, ASC-H, HSIL, atypical glandular cells, or adenocarcinoma in situ, etc.; AND (b) detection of at least 1 of HPV types 31, 33, 45, 52 or 58 by LVPP or EEC swab at the same study visit. Incidence is defined as the number of cases of persistent infection per 10,000 person-years of follow-up in a treatment arm.
Stage I: Geometric Mean Titers of HPV 31, 33, 45, 52 , and 58 Antibodies | 1 Month Post Vaccination 3 (Month 7)
  Serum antibodies to HPV types 31/33/45/52 /58 are measured with cLIA. Titers are reported in milli Merck Units/mL.
Stage I: Percentage of Participants Who Seroconvert by cLIA to HPV Types 31, 33, 45, 52 , and 58 | 1 Month Post Vaccination 3 (Month 7)
  Serum antibody titers for HPV types 31/33/45/52 /58 will be determined using cLIA. The percentage of participants that achieve the serostatus cut-offs for seroconversion for each HPV type will be summarized.
Stage II: Combined Incidence of HPV 31-, 33-, 45-, 52-, and 58-related CIN 1/2/3, AIS, and cervical cancer | Month 7 to Month 90
  This endpoint is defined to have occurred if on a single cervical biopsy, ECC, LEEP or Conization (cold knife/laser) specimen, there is: (a) a pathology panel consensus diagnosis of CIN (Grade 1, 2 or 3), AIS, or cervical cancer; AND (b) detection of at least 1 of HPV types 31, 33, 45, 52 or 58 by Thinsection PCR in an adjacent section from the same tissue block. Disease incidence is defined as the number cases per 10,000 person-years of follow-up in a treatment arm.
Stage II: Combined Incidence of HPV 31-, 33-, 45-, 52-, and 58-related genital warts, CIN 2/3, AIS, cervical cancer, VIN 2/3, VaIN 2/3, vulvar cancer, and vaginal cancer | Month 7 up to Month 90
  This endpoint is defined to have occurred if on a single biopsy or excised tissue, there is: (a) a Pathology Panel consensus diagnosis of CIN (grade 2 or 3), AIS, cervical cancer, VIN (grade 2 or 3), VaIN (grade 2 or 3), vulvar cancer, or vaginal cancer; AND (b) detection of at least 1 of HPV types 31, 33, 45, 52 or 58 by Thinsection PCR in an adjacent section from the same tissue block. Incidence is defined as the number of cases of persistent infection per 10,000 person-years of follow-up in a treatment arm.
Stage II: Combined Incidence of HPV 31-, 33-, 45-, 52-, and 58-related genital warts, CIN 1/2/3, AIS, cervical cancer, VIN 1/2/3, VaIN 1/2/3, vulvar cancer, and vaginal cancer | Month 7 to Month 90
  This endpoint is defined to have occurred if on a single biopsy or excised tissue, there is: (a) a Pathology Panel consensus diagnosis of CIN (grade 1, 2 or 3), AIS, cervical cancer, VIN (grade 1, 2 or 3), VaIN (grade 1, 2 or 3), vulvar cancer, or vaginal cancer; AND (b) detection of at least 1 of HPV types 31, 33, 45, 52 or 58 by Thinsection PCR in an adjacent section from the same tissue block. Disease incidence is defined as the number cases per 10,000 person-years of follow-up in a treatment arm.
Stage II: Combined Incidence of HPV 31-, 33-, 45-, 52- , or 58-related Cervical, Vaginal and External Genital Biopsy and Definitive Therapy | Month 7 up to Month 90
  This endpoint is defined to have occurred if a participant is found to have: (a) a cervical, vaginal or external genital biopsy or definitive therapy; AND (b) a tissue sample from such procedure was detected as PCR positive for at least 1 of HPV types 31, 33, 45, 52 or 58, regardless of the pathology diagnosis of such tissue sample. Incidence of biopsy and definitive therapy will be summarized as the number of cases per 10,000 person-years of follow-up in a treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (6):
- China (6):
  - Lingchuan Center for Disease Control and Prevention ( Site 0002), Guilin, Guangxi
  - Quanzhou Center for Disease Control and Prevention ( Site 0001), Guilin, Guangxi
  - Xiangyuan Center for Disease Control and Prevention ( Site 0003), Changzhi, Shanxi
  - Yanhu Center for Disease Control and Prevention of Yuncheng ( Site 0004), Yuncheng, Shanxi
  - Mianyang Center for Disease Control and Prevention ( Site 0005), Mianyang, Sichuan
  - Santai County Center for Disease Control and Prevention ( Site 0006), Mianyang, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263